CLINICAL TRIAL: NCT05981703
Title: A Phase 1 Study Investigating the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of HPK1 Inhibitor BGB-26808 Alone or in Combination With Anti-PD-1 Monoclonal Antibody Tislelizumab in Patients With Advanced Solid Tumors
Brief Title: A Study Investigating BGB-26808 Alone or in Combination With Tislelizumab in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-26808-101; CTR20240210 (Other: ChinaDrugTrials)
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumor; Solid Tumor
Keywords: advanced solid tumor; BGB-26808; BGB-A317; Tislelizumab; PD1; HPK1
MeSH Terms: interventions — tislelizumab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1a: Dose Escalation (Experimental): Sequential cohorts of increasing dose levels of BGB-26808 will be evaluated as monotherapy and in combination with tislelizumab.
  Interventions: Drug: BGB-26808; Drug: Tislelizumab
- Phase 1b: Dose Expansion (Experimental): Recommended doses for expansion (RDFEs) for BGB-26808 from Phase 1a in combination with tislelizumab plus chemotherapy will be evaluated.
  Interventions: Drug: BGB-26808; Drug: Tislelizumab; Drug: Chemotherapy

INTERVENTIONS:
Drug: BGB-26808 — Planned doses administered orally as a tablet daily.
Drug: Tislelizumab — Planned doses administered by intravenous infusion.
  Other Names: BGB-A317
Drug: Chemotherapy — Administered in accordance with relevant local guidelines and/or prescribing information.
  Arms: Phase 1b: Dose Expansion

SUMMARY:
This is an open-label, multicenter, and nonrandomized dose escalation and dose expansion study to evaluate BGB-26808 as monotherapy or in combination with tislelizumab in participants with advanced solid tumors. The main purpose of this study is to explore the recommended dosing for BGB-26808.

DETAILED DESCRIPTION:
Our company, previously known as BeiGene, is now officially BeOne Medicines. Because some of our older studies were sponsored under the name BeiGene, you may see both names used for this study on this website.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide a signed and dated written informed consent prior to any study-specific procedures, sampling, or data collection.
2. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1.
3. Phase 1a: Participants with histologically or cytologically confirmed advanced, metastatic, and unresectable solid tumors that are immune-sensitive who have previously received standard systemic therapy, or for whom treatment is not available or not tolerated, or for whom treatment is determined not appropriate based on investigator's judgment and who have not received prior therapy targeting hematopoietic progenitor kinase 1 (HPK1).
4. Phase 1b: Participants with histologically confirmed locally advanced unresectable or metastatic tumor types and who have not had prior systemic treatment. Participants who received prior systemic therapy in a neo-adjuvant or adjuvant setting with curative intent for nonmetastatic disease must have experienced a disease-free interval of ≥ 6 months from the last dose of systemic therapy prior to the first dose of study treatments.
5. ≥ 1 measurable lesion per RECIST v1.1.
6. Able to provide an archived tumor tissue sample.
7. Adequate organ function.
8. Females of childbearing potential must be willing to use a highly effective method of birth control for the duration of the study, and for ≥ 90 days after the last dose of BGB-26808, or for ≥ 120 days after the last dose of tislelizumab, or for ≥ 180 days after the last dose of chemotherapy.
9. Nonsterile males must be willing to use a highly effective method of birth control for the duration of the study treatment period and for ≥ 90 days after the last dose of BGB-26808, or for ≥ 120 days after the last dose of tislelizumab, or for ≥ 180 days after the last dose of chemotherapy.

Exclusion Criteria:

1. Prior treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-TIGIT, anti-CTLA4, or any other antibody or drug specifically targeting T-cell costimulation or checkpoint pathways.
2. Uncontrollable pleural effusion, pericardial effusion, or ascites requiring frequent drainage or medical intervention.
3. Clinically significant bleeding from the gastrointestinal tract within 28 days before the first dose of study treatment(s).
4. Active leptomeningeal disease or uncontrolled, untreated brain metastasis.
5. Active autoimmune diseases or history of autoimmune diseases that may relapse
6. Any malignancy ≤ 3 years before the first dose of study treatment(s) except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated with curative intent (eg, resected basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix or breast).
7. Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤ 14 days before the first dose of study treatment(s).
8. History of interstitial lung disease, noninfectious pneumonitis, or uncontrolled lung diseases including pulmonary fibrosis, acute lung diseases.
9. Uncontrolled diabetes.
10. Infection (including tuberculosis infection) requiring systemic (oral or intravenous) antibacterial, antifungal, or antiviral therapy ≤ 14 days before the first dose of study treatment(s).

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From the first dose of study drug(s) to 90 days after the last dose or initiation of a new anticancer therapy, whichever occurs first; up to approximately 12 months
  Number of participants with AEs and SAEs, including findings from physical examinations, electrocardiograms (ECGs), laboratory assessments, and that meet protocol-defined dose-limiting toxicity criteria.
Phase 1a: Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD) of BGB-26808 | Approximately 1 month
  MTD is defined as the highest dose evaluated for which estimated toxicity rate is the closest to the target toxicity rate. MAD is defined as the highest dose administered if MTD is not reached.
Phase 1a: Recommended Dose for Expansion (RDFE) of BGB-26808 | Approximately 1 month
  RDFE of BGB-26808 alone or in combination with tislelizumab will be determined based upon the MTD or MAD.
Phase 1b: Overall Response Rate (ORR) | Approximately 6 months
  ORR is defined as the percentage of participants who had confirmed complete response (CR) or partial response (PR) assessed by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

SECONDARY OUTCOMES:
Phase 1a: ORR | Approximately 6 months
  ORR is defined as the percentage of participants who had confirmed complete response (CR) or partial response (PR) assessed by the investigator using RECIST v1.1.
Phase 1a and 1b: Duration of Response (DOR) | Approximately 9 months
  DOR is defined as the time from the first determination of an objective response per RECIST v1.1 until the first documentation of disease progression or death, whichever occurs first as assessed by the investigator.
Phase 1a and 1b: Disease Control Rate (DCR) | Approximately 6 months
  DCR is defined as the percentage of participants with best overall response of CR, PR, or stable disease. It will be summarized similarly as ORR as assessed by the investigator.
Phase 1a and 1b: Clinical Benefit Rate (CBR) | Approximately 6 months
  CBR is defined as the percentage of participants with best overall response of confirmed CR, PR, or stable disease lasting ≥ 24 weeks as assessed by investigator.
Phase 1b: Progression Free Survival (PFS) | Approximately 9 months
  PFS is defined as the time from the date of the first dose of study drug(s) to the date of the first documentation of progressive disease assessed by the investigator using RECIST v1.1 or death, whichever occurs first.
Phase 1a: Maximum observed plasma concentration (Cmax) for BGB-26808 | Approximately 1 month
Phase 1a: Minimum observed plasma concentration (Cmin) for BGB-26808 | Approximately 6 months
Phase 1a: Time to maximum plasma concentration (Tmax) for BGB-26808 | Approximately 1 month
  Pharmacokinetic analysis for BGB-26808 concentrations, alone or in combination with tislelizumab. Single-dose and steady-state PK parameters.
Phase 1a: Half-life (t1/2) for BGB-26808 | Approximately 1 month
Phase 1a: Area under the concentration-time curve (AUC) for BGB-26808 | Approximately 2 months
Phase 1a: Apparent clearance (CL/F) for BGB-26808 | Approximately 1 month
Phase 1a: Apparent volume of distribution (Vz/F) for BGB-26808 | Approximately 1 month
Phase 1a: Accumulation ratio for BGB-26808 | Approximately 2 months
Phase 1b: Plasma concentrations of BGB-26808 | Approximately 2 months
Phase 1b: Number of Participants with AEs and SAEs | From the first dose of study drug(s) to 90 days after the last dose or initiation of a new anticancer therapy, whichever occurs first; up to approximately 12 months
  Number of participants with AEs and SAEs, including findings from physical examinations, ECGs, laboratory assessments, and that meet protocol-defined dose-limiting toxicity criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeOne Medicines
Locations (26):
- United States (8):
  - City of Hope National Medical Center, Duarte, California
  - University of Southern Californianorris Comprehensive, Los Angeles, California
  - Yale University, Yale Cancer Center, New Haven, Connecticut
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - John Theurer Cancer Center Hackensack University Medical Center, Hackensack, New Jersey
  - Icahn School of Medicine At Mount Sinai, New York, New York
  - Providence Portland Medical Center, Portland, Oregon
  - The University of Texas Md Anderson Cancer Center, Houston, Texas
- Australia (4):
  - Southside Cancer Care, Miranda, New South Wales
  - Macquarie University, North Ryde, New South Wales
  - Icon Cancer Centre Kurralta Park, Kurralta Park, South Australia
  - Linear Clinical Research, Nedlands, Western Australia
- China (12):
  - The First Affiliated Hospital of Anhui Medical Universitygaoxin Branch, Hefei, Anhui
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Tongji Hospital,Tongji Medical College of Hustsino French New City Branch, Wuhan, Hubei
  - The First Hospital of China Medical University Hunnan Branch, Shenyang, Liaoning
  - Jining No Peoples Hospital West Branch, Jining, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Shanghai East Hospital Branch Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Sichuan Academy of Medical Sciences and Sichuan Provincial Peoples Hospital, Chengdu, Sichuan
  - Hangzhou First Peoples Hospital, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province (East), Taizhou, Zhejiang
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Harbour Cancer and Wellness, Auckland

IPD SHARING:
Plan to Share IPD: Yes
BeOne shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeOne shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeOne review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beonemedicines.com/science/clinical-trials/